CLINICAL TRIAL: NCT07272473
Title: Effects of Cervical Mobilization on Dizziness, Balance, and Joint Position Sense in Patients With Meniere's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, ASSOCIATE PROFESSOR, Abant Izzet Baysal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AIBU-FTR-OOP-10
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Meniere Disease
Keywords: Endolymphatic hydrops; Postural Balance; Tinnitus; Position Sense; Kinesthesis; Vestibular Sense; Neck Pains
MeSH Terms: conditions — Meniere Disease; Endolymphatic Hydrops; Tinnitus; Neck Pain

STUDY DESIGN:
Intervention Model Description: There will be a total of 3 groups in the study, two intervention groups and one control group. All groups will continue their routine betahistine treatment. The control group will receive only this standard therapy. Intervention group 1 will receive an additional intervention consisting of 20 minutes of vestibular rehabilitation and 10 minutes of cervical mobilization. Intervention group 2 will receive an additional total of 30 minutes of vestibular rehabilitation. A total of 33 people, 11 in each group, will be included in the study.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vestibular Rehabilitation + Cervical Mobilization (Experimental): Participants receive both vestibular rehabilitation and cervical mobilization interventions.
  Interventions: Other: Vestibular Rehabilitation + Cervical Mobilization
- Vestibular Rehabilitation Alone (Active Comparator): Participants receive vestibular rehabilitation only, administered for 30 minutes per session, twice a week for 6 weeks.The program will include adaptation exercises, habituation exercises, and compensation exercises.
  Interventions: Other: vestibular rehabilitation
- Control Group (No Intervention): Participants receive standard therapy only and do not receive vestibular rehabilitation or cervical mobilisation.

INTERVENTIONS:
Other: Vestibular Rehabilitation + Cervical Mobilization — Treatment will be administered twice a week for 6 weeks, consisting of 20 minutes of vestibular rehabilitation and 10 minutes of cervical mobilization, each lasting 30 minutes. Vestibular rehabilitation will include adaptation exercises, habituation exercises, and compensation exercises. For cervical mobilization, participants will first undergo 3-4 minutes of suboccipital relaxation while lying supine to help them relax, then 2-3 minutes of cervical traction will be applied, and then, while sitting, they will mobilize the C1 and C2 vertebrae using the Mulligan concept.
  Arms: Vestibular Rehabilitation + Cervical Mobilization
Other: vestibular rehabilitation — Vestibular rehabilitation will be applied for 30 minutes, twice a week, for 6 weeks. Adaptation exercises, habituation exercises, and compensation exercises will be applied as vestibular rehabilitation.
  Arms: Vestibular Rehabilitation Alone

SUMMARY:
The study will employ a stratified randomization method. Patients presenting to the Afyonkarahisar Health Sciences University Health Application and Research Center, Ear, Nose, and Throat Outpatient Clinic, with a definitive diagnosis of Meniere's disease, unilateral or bilateral involvement, and who consent to participate in the study will be divided into three groups. The control group will receive only their routine Betahistine. Their usual treatment will remain unchanged. The first study group will receive 20 minutes of Vestibular Rehabilitation (VR) and 10 minutes of cervical mobilization in addition to their routine Betahistine. The second study group will receive 30 minutes of VR in addition to Betahistine. The study will last 6 weeks. Participants will be assessed using a sociodemographic information questionnaire, the Dizziness Handicap Inventory (DHI), the Vertigo Symptom Scale (VSS), the Neck Disability Index (NDI), the International Tinnitus Inventory (ITI), balance assessment with the K-Force Plates, and joint position sense and proprioception assessment with the Kinvent Physio K-Move. All assessments will be conducted twice, before and after treatment.

DETAILED DESCRIPTION:
Patients who have been diagnosed with Meniere's disease and who have applied to the Afyonkarahisar Health Sciences University Health Practice and Research Center, Ear, Nose, and Throat Outpatient Clinic will be included in the study.

The study will employ a stratified randomization method. Patients who have been diagnosed with Meniere's disease and have unilateral or bilateral involvement and who agree to participate in the study will be divided into three groups. The control group will only receive their routine Betahistine. Their usual treatments will remain unchanged. The first study group will receive 20 minutes of Vestibular Rehabilitation (VR) and 10 minutes of cervical mobilization in addition to their routine Betahistine. The second study group will receive 30 minutes of VR in addition to Betahistine. The study will last 6 weeks. During the VR sessions:

1. Adaptation exercises
2. Habituation exercises
3. Compensation exercises. A 6-week exercise protocol will be developed. The exercises will gradually increase in difficulty each week. Adaptation exercises will include visual tracking of a moving object while the head is stationary, and tracking objects in different directions while walking. Habituation exercises will include challenging exercises such as coming from lying down to sitting quickly and rising from sitting to standing. Compensation exercises will include walking on surfaces of varying hardness, standing on a balance board, and balancing on a trampoline, each with increasing difficulty each week.

For cervical mobilization, participants will first undergo 3-4 minutes of suboccipital release while lying on their backs to relax, then 2-3 minutes of cervical traction will be applied, and then, while sitting, they will mobilize the C1 and C2 vertebrae using the Mulligan concept.

Participants will be assessed using a sociodemographic questionnaire, the The Dizziness Handicap Inventory (DHI), the Vertigo Symptom Scale (VSS), the Neck Disability Index (NDI), the International Tinnitus Inventory (ITI), balance assessment with the K-Force Plates, and joint position sense and proprioception assessment with the Kinvent Physio K-Move. All assessments will be conducted twice: at baseline and after 6 weeks. This will allow for comparison of the three groups and provide a pre- and post-treatment assessment.

ELIGIBILITY:
Inclusion Criteria:

* Definitive clinical diagnosis of unilateral or bilateral Meniere's disease
* Age between 18 and 60 years
* Presence of fluctuating symptoms or chronic imbalance for at least 3 months
* Cognitive ability to participate in balance rehabilitation tasks (Mini Mental State Examination score ≥ 24)
* Willingness to participate in the study and provide informed consent

Exclusion Criteria:

* Diagnosis of vertigo not associated with Meniere's disease
* Presence of another acute medical condition
* Neurological, psychological, or cognitive dysfunction
* History of orthopedic surgery within the last 3 months
* Planned surgical intervention during the rehabilitation program
* Cervical spine instability
* Acute cervical trauma
* Vertebral artery insufficiency

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-20 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-05-05 (Estimated)

PRIMARY OUTCOMES:
Balance assessments | From enrollment to the end of treatment at 6 weeks
  Balance assessments will be conducted statically and dynamically using K-Force Plates. Both bilateral and unilateral balance tests will be conducted for static balance assessments. In the bilateral balance test, participants will be tested on both feet, first with their eyes open and then with their eyes closed. In the unilateral test, participants will first be asked to stand on their right and left legs for 10 seconds, with their eyes open, and then three repetitions, with the average calculated. They will then be asked to stand on their right and left legs, again, with their eyes closed.
  In the dynamic balance test, participants will be asked to jump and descend from a step placed 19 cm above the force plate. (Both feet will be suspended before landing.) They will then be asked to balance with their hands on their hips for 15 seconds. If the participant moves their foot or loses their balance completely, the trial will be cancelled and repeated.

SECONDARY OUTCOMES:
Dizziness assesment | From enrollment to the end of treatment at 6 weeks
  The Dizziness Handicap Inventory (DHI) will be used to assess dizziness. DHI was developed by Jacobson and Newman in 1990. The DHI consists of 25 items that identify factors that aggravate dizziness and balance disorders in patients, as well as the sensory and functional consequences of vestibular system disorders. Sub-inventories are designed to determine the physical, sensory, and functional effects of vestibular system disorders.
  Each question has a yes (4 points), no (0 points), and sometimes (2) response. When scoring the sub-items of the inventory, a score of 28 is recommended as the threshold for determining physical disability, and a score of 36 is recommended as the threshold for determining functional and sensory disability. High scores are interpreted as indicating that the patient's dizziness complaint significantly impedes their life. The Turkish validity and reliability test of the inventory was conducted.
Vertigo Symptom Assesment | From enrollment to the end of treatment at 6 weeks
  The Vertigo Symptom Scale (VSS) is used to assess the frequency of symptoms such as imbalance, somatic symptoms, autonomic symptoms, anxiety, and panic, which are commonly encountered in patients with vertigo and feelings of imbalance. The scale consists of two subsections: the Vertigo Symptom Scale-Vertigo Section (VSS-V), which relates to vertigo and balance disorders, and the Vertigo Symptom Scale-Anxiety Section, which relates to autonomic disorders and anxiety symptoms. The VSS-V consists of 8 questions (0-32 points), and the VSS-A consists of 7 questions (0-28 points). Symptom frequency is scored from 0= never, 1= very infrequently, 2= often, 3= often (every week), and 4= very often (more than 1 day per week on average). Patients are asked to answer these questions about their dizziness, thinking back to the past month. Higher scores (maximum 60) indicate an increased frequency of experiencing vertigo-related symptoms. A score of ≥12 is defined as severe dizziness.
Neck Disability Assessment | From enrollment to the end of treatment at 6 weeks
  The Neck Disability Index (NDI) is a 10-item assessment tool covering pain severity, personal care, weightlifting, reading, headache, concentration, working, driving, sleep, and rest. It measures the level of functional limitations associated with the neck. Each item is scored from 0 (no disability) to 5 (maximum disability). The highest total score is 50. It is accepted that as an individual's score increases, the level of disability due to neck pain also increases. A total score of 0 indicates no disability, while a score of 50 indicates maximum disability. According to the assessment, scores between 0 and 4 are classified as "no disability", 5-14 as "mild disability", 15-24 as "moderate disability," 25-34 as "severe disability," and 35 and above as "complete disability."
Tinnitus Assessment | From enrollment to the end of treatment at 6 weeks
  The International Tinnitus Inventory (ITI), aims to assess the multidimensional effects of tinnitus on individuals.This assessment encompasses perceptions of hearing, general health status, sleep patterns, inner peace, social relationships, daily living activities, enjoyment of life, and the level of discomfort caused by tinnitus. The inventory consists of eight items, and each item is scored from 1 to 5; the total score ranges from 8 to 40. Lower total scores indicate a greater perception of the negative effects of tinnitus on the individual.
Proprioception Assessment | From enrollment to the end of treatment at 6 weeks
  The Kinvent Physio K-Move device is a wireless, portable motion sensor developed for the objective assessment of movement. This device is used specifically in physiotherapy and rehabilitation processes to precisely measure and monitor joint range of motion (ROM) and joint position sense. Validity and reliability of the device for assessing joint position sense and proprioception have been established.
  The device measures head flexion, extension, lateral flexion, and rotation angles. During the measurements, participants' cervical joint range of motion will be assessed first. Participants will be seated in a comfortable sitting position with their feet flat on the floor and their heads in a neutral position, arms at their sides. Participants will be instructed and demonstrated on all movements they will perform before the assessment.

CONTACTS AND LOCATIONS:
Overall Officials: omer pala, associate professor, Study Director — Abant Izzet Baysal University
Locations (1):
- Afyonkarahisar Health Sciences University Health Application and Research Center, Ear, Nose and Throat Polyclinic, Afyonkarahisar, Afyonkarahisar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No